CLINICAL TRIAL: NCT02853266
Title: Measurement of Antibodies in Adults With a History of Kawasaki Disease
Acronym: KAWASAKI Ac
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0477
Record Dates: First submitted 2016-07-21; First posted 2016-08-02 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Kawasaki Disease
Keywords: Kawasaki disease; non-cruzi-related antibody (NCRA)
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — de-identified and study coded serum sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients KD: adults with a history of KD in childhood
  Interventions: Other: laboratory biomarker analysis
- control group: healthy adults volunteers
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Archived serum samples are analysed for measurement of biomarker NCRA

SUMMARY:
Kawasaki disease (KD) is an acute systemic vasculitic syndrome with coronary tropism. It has been reported worldwide, but it is ten times more common in Asian population. It is the second vasculitis of the child by its frequency after rheumatoid purpura. It occurs in 80% of cases between 1 and 5 years, with a maximal incidence around the age of 12 months.

KD is not well understood and the cause is yet unknown. It may be an autoimmune disorder. The problem affects the mucous membranes, lymph nodes, walls of the blood vessels, and the heart.The clinical picture of KD associate a persistent fever and an antipyretics resistance with mucocutaneous signs and bulky cervical lymphadenopathy usually unilateral.

There is currently no vaccine available against Kawasaki disease so it is extremely important to be able to recognize symptoms before they set in and become too severe.

Chagas disease (CD) is caused by the parasite Trypanosoma cruzi. Acute CD occurs immediately after infection, may last up to a few weeks or months. Infection may be mild or asymptomatic. There may be fever or swelling around the site of inoculation, and acute infection may result in severe inflammation of the heart muscle. The notion that the pathology of CD has an autoimmune component was initially based on the finding of circulating antibodies binding heart tissue antigens in patients chronically infected with T. cruzi.

A recent study reports a possible antigen (non-cruzi-related antibody NCRA) mimicry characterized by a serological reactivity to a well-defined T. cruzi antigen in blood samples from individuals not exposed to the parasite. The measured seroprevalence of such cross-reactivity is in favor of a highly prevalent immunogen acquired in childhood.

There are similarities in mechanism of CD and KD: it could be interesting to explore the presence of NCRA in blood samples from adults with a history of KD.

The objective of the study is the measurement of the biomarker NCRA in serum in adults with a history of KD compare to a control population. This measurement and the prevalence may permit to associate the NCRA to a possible pathogenic agent.

ELIGIBILITY:
Inclusion Criteria:

* History of KD before the age of 18, with or without macroscopic coronary lesions in the childhood phase. (KD group only)
* 18 years old or older at the time of the study.
* Agree on participating to all explorations of the study.
* Accept genotyping.
* Absence of cardiovascular risk factors

Exclusion Criteria:

* - Atypical KD (KD group only)
* Documented or suspected coronary ischemia,
* Refusal to participate to the study or sign the consent
* Contra-indication to the injection of iodinated contrast agents (allergy, renal failure)
* Hypersensitivity to dobutamine,
* No effective contraception method for females with child bearing potential,
* Breastfeeding, or pregnant females,
* Treatment modifying endothelial reactivity
* History of severe intolerance to iodinated contrast agents,
* Subjects who can't hold their breath for at least 20 seconds,
* Irregular or absence of sinus rhythm, especially atrial or ventricular arrhythmia
* Unability to give information to the subject,
* No coverage from a Social Security system
* Deprivation of civil rights

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients enrolled in Kawasaki study
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2011-09; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of NCRA in the KD population vs control population. | at recruitment time. (Day 0)
NCRA concentration in the KD population vs control population. | at recruitment time. (Day 0)
  Measurement of the biomarker NCRA in serum in adults with a history of KD vs control population

CONTACTS AND LOCATIONS:
Overall Officials: François Gueyffier, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Louis Pradel - Service de Pharmacologie Clinique, Bron, France